CLINICAL TRIAL: NCT07236918
Title: The Concert Therapy: An Arts-Based Pilot Study on Music, Breathing, and Movement for Stress Reduction and Wellbeing
Brief Title: The Concert Therapy Pilot Study for Stress Reduction and Wellbeing
Acronym: TCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BeHnam KhodaRahmi (Industry)
Responsible Party: Sponsor-Investigator, BeHnam KhodaRahmi, Founder & Principle Investigator, The Concert Therapy
Organization: The Concert Therapy (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TCT-BKH-2025-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Stress Reduction; Psychological Wellbeing; Mental Health; Music Therapy
Keywords: The Concert Therapy; music therapy; arts-based intervention; breathing exercises; movement; stress; wellbeing; mental health; mindfulness; relaxation; live performance; pilot study
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two parallel cohorts receive the same arts-based intervention delivered via different formats: one in-person and one online. Pre-post within-group changes are evaluated.
Masking Description: Open-label study; no masking applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person The Concert Therapy Session (Experimental): Single-session arts-based intervention delivered in person, combining live music, guided breathing, and gentle movement in a structured three-part format (calming music, breathing & movement, uplifting music).
  Interventions: Behavioral: The Concert Therapy
- Online The Concert Therapy Session (Experimental): Single-session arts-based intervention delivered online through a live, interactive platform, featuring the same music, breathing, and movement structure as the in-person session.
  Interventions: Behavioral: The Concert Therapy

INTERVENTIONS:
Behavioral: The Concert Therapy — The Concert Therapy is an arts-based behavioural intervention integrating live music, guided breathing, and gentle movement. Each session follows a three-part structure designed to promote relaxation, body awareness, and emotional well-being through synchronised rhythm and breath.
  Participants take part in a single session, delivered either in person (approximately 66 minutes) or online (approximately 33 minutes), depending on their assigned group. Both formats use live, interactive facilitation and follow the same sequence of musical and breathing exercises adapted to the delivery mode.

SUMMARY:
The Concert Therapy is an arts-based, pilot interventional study designed to explore the effects of live music, guided breathing, and movement on stress reduction and overall wellbeing. Participants take part in one in-person session and one online session integrating musical performance, collective breathing rhythms, and body awareness techniques. The study aims to evaluate pre- and post-intervention changes in perceived stress and emotional wellbeing among adult participants.

DETAILED DESCRIPTION:
This pilot study investigates the effects of The Concert Therapy, an arts-based, multi-sensory approach combining music, guided breathing, and mindful movement, on stress reduction and wellbeing.

The intervention includes two formats: one in-person session and one online session delivered via a live, interactive platform. Each session features structured breathing exercises, live musical interaction, and guided movement sequences designed to synchronize rhythm, breath, and body awareness.

A pre-post design is used, with data collected immediately before and after both sessions. Quantitative outcomes include changes in the Perceived Stress Scale (PSS-10), while qualitative data will be gathered through open-ended feedback regarding participants' emotional, physical, and social experiences.

The study aims to generate preliminary evidence on the feasibility and potential benefits of The Concert Therapy as an accessible, arts-based intervention for stress management and wellbeing in both physical and virtual settings.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older.

* Able to understand and provide informed consent.
* Willing and able to participate in a 60-minute in-person or 33-minute online session of The Concert Therapy.
* Able to complete brief questionnaires in English before and after the session.

Exclusion Criteria:

* Self-reported severe mental health conditions requiring medical treatment.
* Significant hearing impairment that would limit engagement with music.
* Inability to access the online platform (for online participants).
* Previous participation in The Concert Therapy study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2025-11-16 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS-10) Score | Pre-session to immediately post-session (same day)
  Change in participants' perceived stress levels measured by the 10-item Perceived Stress Scale (PSS-10) before and immediately after participation in The Concert Therapy session (in-person or online). Higher scores indicate greater stress.

SECONDARY OUTCOMES:
Participant Feedback on Emotional and Physical Well-being | Immediately post-session
  Qualitative feedback collected after The Concert Therapy session, exploring participants' experiences of calmness, relaxation, enjoyment, and social connectedness. Responses will be analysed thematically.

CONTACTS AND LOCATIONS:
Locations (1):
- The Concert Therapy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared; only aggregated, de-identified results will be published.

REFERENCES:
- See also: Related Info — https://www.theconcerttherapy.com